CLINICAL TRIAL: NCT07211269
Title: Individual Differences in Cognitive Control Predict Real-time fMRI Neurofeedback Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Shuxia Yao, Dr, University of Electronic Science and Technology of China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-95
Record Dates: First submitted 2025-08-28; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Neurofeedback Performance; Interoception; Cognitive Control

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurofeedback group (Experimental): Participants received real-time neurofeedback information from the target regulation brain region.
  Interventions: Other: Real-time fMRI neurofeedback training

INTERVENTIONS:
Other: Real-time fMRI neurofeedback training — Real-time neurofeedback information is computed using the Turbo Brain voyager (TBV) 4.0 software (Brain Innovation, Maastricht, The Netherlands). Functional images are collected and processed in real time based on contrasts of regulation vs. rest conditions. The BOLD signal of the target region is then transformed into visual bars and displayed to participants via the projector screen while participants keep using regulation strategy (heartbeat interoception in our study) to upregulate the target region.

SUMMARY:
The goal of this study is to investgate whether individual differences of cognitive control capacity could predict neurofeedback performance and the behavioral effects resulting from successful anterior insula regulation via interoceptive strategy.

DETAILED DESCRIPTION:
The experimental protocol comprises two visits with a 3-7 days interval. The first visit includes: (1) completion of standardized psychological questionnaires, (2) pre-test of the heartbeat counting task (HCT), and (3) four validated cognitive control tasks, including the Go/No-Go task, Stroop task, Task-switching task, N-back task. The main task of the second visit is a fMRI task followed by a post-test of the HCT. The MRI scanning protocol includes anatomical scan, two resting-state scans (pre- and post-training), four runs of fMRI neurofeedback training and a transfer run without feedback. During the regulation block of the training task, participants are asked to upregulate the anterior insula activity followed by a pain empathy rating and strategy efficacy rating. All participants receive real-time neurofeedback from the left anterior insula. Scores of questionnaires including Positive and Negative Affect Schedule, Beck Depression Inventory-Ⅱ, Autism Spectrum Quotient, State-Trait Anxiety Inventory, Interpersonal Reactivity Index, Toronto Alexithymia scale, Bermond-Vorst Alexithymia Questionnaire, Interoceptive Confusion Questionnaire, Multidimensional Assessment of Interoceptive Awareness, Cognitive Flexibility Inventory are also collected before the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any past or present psychiatric or neurological disorders

Exclusion Criteria:

* History of brain injury Medical or mental illness and color blindness or weakness.
* The presence of metal in the body or claustrophobia.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2025-12-27 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
BOLD signal of the anterior insula during neurofeedback training | 1 hour
  The anterior insula activity induced by regulation relative to rest blocks in the neurofeedback training task and transfer task.
Behavioral measurements in the cognitive control tasks | 1 hour
  Response time and accuracy are recorded in the cognitive control tasks (i.e., the Go/No-Go task, Stroop task, Task-switching, N-back task).

SECONDARY OUTCOMES:
Pain empathy ratings scores | 1 hour
  Subjects were required to rate their empathic feeling towards painful pictures on a Likert Scale ranging from 1-9 (1 = not at all and 9 = very painful) after each block.
Strategy efficacy rating scores | 1 hour
  Subjects were required to rate the strategy efficacy on a Likert Scale ranging from 1-9 (1 = not at all and 9 = very) after each block.
Intero-ceptive accuracy | 15 minutes
  The ratio of participants' perceived number of heartbeat relative to the recorded number of heartbeat in the heartbeat counting task.
Confidence rating scores of interoceptive sensitivity | 15 minutes
  Subjects were asked to rate to what extent they can feel their heartbeat based on a Likert Scale ranging from 1-9 (1 = very low and 9 = very high) in the heartbeat counting task.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Shuxia, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Chengdu, China